CLINICAL TRIAL: NCT02293824
Title: Effect of Feedings on Caffeine Pharmacokinetics and Metabolism in Premature Infants
Brief Title: Effect of Feedings on Caffeine in Premature Infants
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00058253
Record Dates: First submitted 2014-11-14; First posted 2014-11-18 (Estimated); Last update posted 2017-09-13 (Actual); Status verified 2017-06

CONDITIONS: Apnea of Prematurity; Premature Newborn; Caffeine
Keywords: Infant, Premature; Caffeine; Pharmacokinetics; Metabolism
MeSH Terms: conditions — Apnea; Premature Birth | interventions — Caffeine; caffeine citrate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Premature infants: Premature infants <29 weeks birth gestational age receiving caffeine per standard of care for the prevention or treatment of apnea of prematurity.
  Interventions: Drug: Caffeine

INTERVENTIONS:
Drug: Caffeine — Given per standard of care.
  Other Names: Caffeine Citrate; Cafcit

SUMMARY:
Almost all infants born <29 weeks gestational age develop apnea of prematurity and are treated with caffeine. Type of diet and disease states may be significant contributors of variability in caffeine metabolism and pharmacokinetics (PK) in this population. This prospective, observational, open-label, opportunistic PK study will compare the population PK of caffeine between infants fed formula and infants fed exclusively breast milk; compare the activities of caffeine metabolizing enzymes between infants fed formula and infants fed exclusively breast milk; and determine the effect of hypoxia, hypotension, and infection on caffeine PK and metabolism in premature infants.

DETAILED DESCRIPTION:
This study will use a consecutive patient sampling approach. All eligible participants admitted at each site will be approached. Caffeine and feedings will be administered per standard of care. Manipulations of caffeine dosing or feeding regimens will not be a part of this protocol. To minimize the amount of blood sampling, the investigators will use a sparse sampling methodology. Urine will be collected for analysis of caffeine and caffeine metabolite concentrations. Caffeine pharmacokinetics will be described by population pharmacokinetic analysis. Urinary concentrations of caffeine and its metabolites will be used to calculate metabolic ratios as markers of enzyme activity.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent from parent(s) or legal guardian(s)
* <29 weeks birth gestational age
* Postnatal age ≤15 days
* Receiving caffeine (intravenous or oral) per standard of care for prevention or treatment of apnea of prematurity

Exclusion Criteria:

* Known major congenital or chromosomal anomaly

Max Age: 15 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Premature infants given caffeine for the prevention or treatment of apnea of prematurity.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2014-12; Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Clearance (CL) of caffeine at steady state | Study days 0, 15, 30, 45, and 60.
  Using population pharmacokinetic analyses

SECONDARY OUTCOMES:
Volume of distribution (V) of caffeine at steady state | Study days 0, 15, 30, 45, and 60
  Using population pharmacokinetic analyses
Caffeine metabolizing enzyme activity using urinary metabolic ratios | Study days 0, 15, 30, 45, and 60
  Activity levels of CYP1A2, xanthine oxidase, and N-acetyltransferase 2
Fold change in caffeine clearance due to hypoxia, hypotension, and infections | Study days 0, 15, 30, 45, and 60
  Effect of hypoxia, hypotension, and infections on caffeine clearance

CONTACTS AND LOCATIONS:
Overall Officials: Phillip B Smith, MD, MPH, MHS, Principal Investigator — Duke Clinical Research Institute
Locations (2):
- United States (2):
  - North Carolina Children's Hospital, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: Undecided
Will consider on a case-by-case basis (de-identified data only)

REFERENCES:
- [Background] Zhao J, Gonzalez F, Mu D. Apnea of prematurity: from cause to treatment. Eur J Pediatr. 2011 Sep;170(9):1097-105. doi: 10.1007/s00431-011-1409-6. Epub 2011 Feb 8. PMID 21301866
- [Background] Di Fiore JM, Bloom JN, Orge F, Schutt A, Schluchter M, Cheruvu VK, Walsh M, Finer N, Martin RJ. A higher incidence of intermittent hypoxemic episodes is associated with severe retinopathy of prematurity. J Pediatr. 2010 Jul;157(1):69-73. doi: 10.1016/j.jpeds.2010.01.046. Epub 2010 Mar 20. PMID 20304417
- [Background] Janvier A, Khairy M, Kokkotis A, Cormier C, Messmer D, Barrington KJ. Apnea is associated with neurodevelopmental impairment in very low birth weight infants. J Perinatol. 2004 Dec;24(12):763-8. doi: 10.1038/sj.jp.7211182. PMID 15329741
- [Background] Clark RH, Bloom BT, Spitzer AR, Gerstmann DR. Reported medication use in the neonatal intensive care unit: data from a large national data set. Pediatrics. 2006 Jun;117(6):1979-87. doi: 10.1542/peds.2005-1707. PMID 16740839
- [Background] Gal P. Caffeine Therapeutic Drug Monitoring Is Necessary and Cost-effective. J Pediatr Pharmacol Ther. 2007 Oct;12(4):212-5. doi: 10.5863/1551-6776-12.4.212. No abstract available. PMID 23055855
- [Background] Blake MJ, Abdel-Rahman SM, Pearce RE, Leeder JS, Kearns GL. Effect of diet on the development of drug metabolism by cytochrome P-450 enzymes in healthy infants. Pediatr Res. 2006 Dec;60(6):717-23. doi: 10.1203/01.pdr.0000245909.74166.00. Epub 2006 Oct 25. PMID 17065585
- [Background] Le Guennec JC, Billon B. Delay in caffeine elimination in breast-fed infants. Pediatrics. 1987 Feb;79(2):264-8. PMID 3808800
- [Background] Xu H, Rajesan R, Harper P, Kim RB, Lonnerdal B, Yang M, Uematsu S, Hutson J, Watson-MacDonell J, Ito S. Induction of cytochrome P450 1A by cow milk-based formula: a comparative study between human milk and formula. Br J Pharmacol. 2005 Sep;146(2):296-305. doi: 10.1038/sj.bjp.0706319. PMID 15997229
- [Background] Supnet MC, David-Cu R, Walther FJ. Plasma xanthine oxidase activity and lipid hydroperoxide levels in preterm infants. Pediatr Res. 1994 Sep;36(3):283-7. doi: 10.1203/00006450-199409000-00003. PMID 7808822
- [Background] Hassoun PM, Yu FS, Cote CG, Zulueta JJ, Sawhney R, Skinner KA, Skinner HB, Parks DA, Lanzillo JJ. Upregulation of xanthine oxidase by lipopolysaccharide, interleukin-1, and hypoxia. Role in acute lung injury. Am J Respir Crit Care Med. 1998 Jul;158(1):299-305. doi: 10.1164/ajrccm.158.1.9709116. PMID 9655743
- See also: Bedford Laboratories. CAFCIT (caffeine citrate) injection, CAFCIT (caffeine citrate) solution. 2013. — http://dailymed.nlm.nih.gov/dailymed/lookup.cfm?setid=fbcd234e-57e1-4da2-a96c-e3f7b7cf6ec0